CLINICAL TRIAL: NCT04258098
Title: Preoperative Mechanical Bowel Preparation With Oral Antibiotics Reduces Surgical Site Infection After Elective Colorectal Surgery for Malignancies: a Propensity Matching Analysis
Brief Title: Prophylatic Effect Preoperative Antibiotics With Mechanical Bowel Preparation in SSIs: A Propensity Analysis
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Prof., Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: OAMBP-02; 2018023 (Other: Sun Yat-sen University 5010 clinical program)
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Surgical Site Infection; Colorectal Cancer
MeSH Terms: conditions — Surgical Wound Infection; Colorectal Neoplasms | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OA+MBP group: Either polyethylene glycol or magnesium sulphate was adopted as laxative one day before surgery. Clyster was conducted on surgery morning. Streptomycin 1g plus metronidazole 0.2g was prescribed 3 times a day for 3 days before surgery in the OA+MBP group patients.
  Interventions: Drug: Oral antibiotics ( Streptomycin ,metronidazole )
- MBP group: Either polyethylene glycol or magnesium sulphate was adopted as laxative one day before surgery. Clyster was conducted on surgery morning. No oral antibiotics was administered to the patients.

INTERVENTIONS:
Drug: Oral antibiotics ( Streptomycin ,metronidazole ) — Either polyethylene glycol or magnesium sulphate was adopted as laxative one day before surgery. Clyster was conducted on surgery morning. Streptomycin 1g plus metronidazole 0.2g was prescribed 3 times a day for 3 days before surgery in the OA+MBP group patients.
  Groups: OA+MBP group

SUMMARY:
Surgical site infections (SSIs) are a major postoperative complication after colorectal surgery. Current study aims to evaluate prophylactic function of oral antibiotic intake (OA) in combination with mechanical bowel preparation (MBP) relative to MBP alone with respect to postoperative SSIs incidence. A retrospective analysis of eligible patients was to conducted using the databases of the Gastrointestinal Surgery Centre, Third Affiliated Hospital of Sun Yat-sen University from 2011 to 2017. Data pertaining to postoperative hospital stay length, expenses, SSIs incidence, anastomotic fistula incidence, and rates of other complications wloud be extracted and compared. A propensity analysis was conducted to minimize bias associated with demographic characteristics.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are a major postoperative complication after abdominal surgery, especially in the colorectal field. With a reported incidence of over 20%, SSIs significantly increase the length of stay (LOS), readmission rate, expenses, and mortality . Therefore, the identification of an effective method of reducing SSIs incidence is critically important.

Colonic bacterial florae are considered to be the major cause of SSIs after elective colorectal procedures, but the most effective means of decreasing this bacterial load remains under debate. Pre-operative mechanical bowel preparation (MBP) was first utilized by surgeons, as it can theoretically remove stool content and associated bacterial load within the bowel and surgical field, thus reducing risk of SSIs. More recently, as antibiotics have come to be widely utilized, the pre-operative administration of un-absorbed oral antibiotics (OA) in combination with MBP was widely conducted.

Multiple trials have been performed to explore the best bowel preparation strategies, but their results remain controversial. Since 2005, several RCTs and meta-analyses have demonstrated MBP alone was not associated with a reduced incidence of SSIs related to patients that did not undergo MBP, whereas MBP patients exhibited paradoxical increases in postoperative ileus, anastomotic leakage, and other complications. Recently, the merit of OA and MBP has been re-discovered in several related retrospective studies which demonstrated a significant decrease in the rate of SSIs.However, as information in these trials was exacted from national databases without any detailed matching between patient groups, the existence of bias in these trials may affect the validity of their results. Furthermore, none of these studies assessed the relative prophylactic effects of the novel MBP mode in right or left-side colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient underwent elective colorectal resection to treat a malignancy;
2. Patient baseline characteristics and operative information were available;
3. MBP (mechanical bowel preparation) was performed before surgery, with or without OA (oral antibiotics).

Exclusion Criteria:

1. Emergency surgery;
2. MBP was not conducted due to ileus or patient refusal;
3. Enough data was not available;
4. Colorectal resection was performed due to benign disease;
5. The procedure was accompanied by other procedures that had the potential to contaminate the incision, such as cholecystectomy or appendectomy;
6. Patients underwent neoadjuvant radiotherapy before surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients were identified by searching the database of the Gastrointestinal Surgery Centre, Third Affiliated Hospital of Sun Yat-sen University from 2011 to 2017.
Sampling Method: Non-Probability Sample
Enrollment: 806 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
SSIs incidence | up to 30 days postoperatively
  Surgical site infection incidence

SECONDARY OUTCOMES:
length of hospital stays | up to 3 months posteroperatively
  length of hospital stays after colorectal surgeries

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lei P, Ruan Y, Yang X, Wu J, Hou Y, Wei H, Chen T. Preoperative mechanical bowel preparation with oral antibiotics reduces surgical site infection after elective colorectal surgery for malignancies: results of a propensity matching analysis. World J Surg Oncol. 2020 Feb 11;18(1):35. doi: 10.1186/s12957-020-1804-4. PMID 32046725